CLINICAL TRIAL: NCT07175974
Title: Effects of a Feldenkrais Method-Based Protocol on Body Fluid Balance and Stress-Related Responses in Healthy Adult Women: A Pilot Study
Brief Title: Feldenkrais Method and Stress-Related Responses in Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Marianna Bellafiore, Professor, University of Palermo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FM-2023-PILOT
Record Dates: First submitted 2025-09-04; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stress, Psychological; Autonomic Nervous System; Hydration; Healthy Volunteers
Keywords: Feldenkrais Method; Mind-Body Intervention; Stress Adaptation; Body Fluid Balance; Psychological Well-Being; Self-Compassion
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either the Feldenkrais Method intervention group or the control group based on availability and willingness to attend all sessions. Outcomes were assessed pre- and post-intervention for both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Feldenkrais Method (Experimental): Participants attended eight consecutive "Awareness Through Movement" (ATM) sessions of the Feldenkrais Method, each lasting 90 minutes, over 8 days (total 12 hours). The protocol focused on improving upper limb functionality, integration with trunk movement, posture, coordination, and body awareness.
  Interventions: Behavioral: Feldenkrais Method - Awareness Through Movement (ATM)
- Control Group - No Intervention (No Intervention): Participants did not receive any intervention or structured physical activity during the 8-day study period. They continued their usual daily routines.

INTERVENTIONS:
Behavioral: Feldenkrais Method - Awareness Through Movement (ATM) — Participants attended eight consecutive sessions of the Feldenkrais Method, each lasting 90 minutes, over 8 days (total 12 hours). Sessions focused on enhancing upper limb functionality, trunk integration, posture, coordination, body awareness, and somatic regulation through slow, mindful, guided movements.
  Arms: Intervention Group - Feldenkrais Method

SUMMARY:
This pilot study aimed to explore whether the Feldenkrais Method, a gentle movement and awareness practice, could help reduce stress and improve well-being in sedentary adult women. Twenty-four women aged 26-59 years were recruited. Participants were assigned to either an intervention group, which completed eight consecutive daily Feldenkrais sessions (90 minutes each), or to a control group.

Before and after the program, all participants were assessed for: resting heart rate (HR), averaged over 5 minutes, and heart rate variability (HRV) to measure nervous system balance; total body water (TBW) and extracellular water (ECW), and a marker of stress response, the Hypothalamic-Pituitary-Adrenal (HPA) axis index, using bioelectrical impedance analysis (BIA); weight and height; and questionnaires to evaluate psychological well-being and self-compassion.

DETAILED DESCRIPTION:
Background and Rationale: The Feldenkrais Method® (FM) is a mind-body approach that uses gentle, slow, and mindful movements to enhance self-awareness, motor control, and movement efficiency. Similar mind-body practices such as Yoga and Tai Chi have been shown to improve autonomic regulation, reduce stress-related biomarkers, and enhance psychological well-being. Chronic stress, particularly in sedentary individuals, can negatively affect the autonomic nervous system (ANS), hypothalamic-pituitary-adrenal (HPA) axis, and cardiovascular health. Despite the growing popularity of FM, evidence regarding its effects on autonomic balance and stress adaptation remains limited.

Study Purpose and Hypothesis: This pilot study aimed to explore whether a short FM-based protocol could influence physiological and psychological responses to stress in healthy adult women. It was hypothesized that participation in an 8-day FM program would improve autonomic regulation, body fluid balance, and psychological well-being.

Study Design: A pilot study was conducted with 24 healthy sedentary women. Participants were assigned to either an intervention group (IG) or a control group (CG) based on their interest and availability to attend all FM sessions. Due to the intensive nature of the intervention and practical constraints, randomization was not performed. All participants provided written informed consent, and the study was approved by the Bioethics Committee of the University of Palermo (Approval No. 129/2023). Assessments were conducted pre- and post-intervention at the "Studio Forte" and the "Functional Assessment Laboratory" of Palermo University between April and July 2023.

Participant Selection and Sedentary Criteria: Inclusion criteria required participants to be healthy, adult sedentary women (≥18 years). Sedentariness was defined according to World Health Organization guidelines: less than 150 minutes per week of moderate-intensity activity, less than 75 minutes per week of vigorous activity, or an equivalent combination. Data were collected using a self-administered questionnaire covering demographic information, education level, occupation, weekly minutes of physical activity, and self-reported medical history.

Intervention: The IG performed eight consecutive Awareness Through Movement (ATM) lessons, each lasting 90 minutes, focusing on upper limb functionality and integration with trunk movements. The CG did not participate in any structured activity during the same period.

Outcome Measures: Physiological outcomes included resting heart rate (HR), averaged over 5 minutes, heart rate variability (HRV) assessed via Polar H10 sensor, total body water (TBW), extracellular water (ECW), and HPA axis index measured through bioelectrical impedance analysis (BIA). Body weight and height were measured by the study operator using a standard digital scale and stadiometer, respectively.

HRV metrics encompassed time-domain (SDNN, RMSSD) and frequency-domain (VLF, LF, HF, LF/HF ratio) parameters. TBW and ECW reflected body fluid distribution, while the HPA axis index provided an indirect measure of neuroendocrine adaptation to stress. The Psychological Well-Being Scale (PWBS) and the Self-Compassion Scale (SCS) were used to assess psychological well-being and self-compassion, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Female (age ≥18 years)
* Healthy (no musculoskeletal disorders or other conditions limiting participation in the Feldenkrais Method protocol)
* Sedentary lifestyle (<150 min/week of moderate-intensity physical activity or <75 min/week of vigorous-intensity activity)

Exclusion Criteria:

* Male
* Presence of acute or chronic medical conditions
* Current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Total Body Water (TBW) | Baseline and post-intervention (8 days)
  Total body water measured via bioelectrical impedance analysis (BIA), in liters (L).
Extracellular Water (ECW) | Baseline and post-intervention (8 days)
  Extracellular water measured via bioelectrical impedance analysis (BIA), in liters (L).
Hypothalamic-Pituitary-Adrenal (HPA) Axis Index | Baseline and post-intervention (8 days)
  Hypothalamic-pituitary-adrenal (HPA) axis index measured via bioelectrical impedance analysis (BIA), expressed as phase angle (PA°).
Resting Heart Rate (HR) | Baseline and post-intervention (8 days)
  Resting heart rate measured using a Polar H10 chest strap, calculated as the average heart rate over a 5-minute period, in beats per minute (bpm).
Standard Deviation of NN intervals (SDNN) | Baseline and post-intervention (8 days)
  SDNN measured from heart rate variability using a Polar H10 chest strap and Kubios HRV software, in milliseconds (ms).
Root Mean Square of Successive Differences (RMSSD) | Baseline and post-intervention (8 days)
  RMSSD measured from heart rate variability using a Polar H10 chest strap and Kubios HRV software, in milliseconds (ms).
Very Low Frequency (VLF) Power | Baseline and post-intervention (8 days)
  VLF power measured from heart rate variability using a Polar H10 chest strap and Kubios HRV software, in milliseconds squared (ms²).
Low Frequency (LF) Power | Baseline and post-intervention (8 days)
  LF power measured from heart rate variability using a Polar H10 chest strap and Kubios HRV software, in milliseconds squared (ms²).
High Frequency (HF) Power | Baseline and post-intervention (8 days)
  HF power measured from heart rate variability using a Polar H10 chest strap and Kubios HRV software, in milliseconds squared (ms²).
LF/HF Ratio | Baseline and post-intervention (8 days)
  LF/HF ratio calculated from heart rate variability using a Polar H10 chest strap and Kubios HRV software (unitless).

SECONDARY OUTCOMES:
Psychological Well-Being Scale (PWBS) | Baseline and post-intervention (8 days)
  Total score on the Psychological Well-Being Scale, in units on a scale.
Self-Compassion Scale (SCS) | Baseline and post-intervention (8 days)
  Total score on the Self-Compassion Scale, in units on a scale.

OTHER OUTCOMES:
Weight | Baseline and post-intervention (8 days)
  Weight measured by the study operator using a standard digital scale, in kilograms (kg).
Height | Baseline and post-intervention (8 days)
  Height measured by the study operator using a stadiometer, in centimeters (cm).

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Exercise Sciences Research Unit, Department of Psychology, Educational Science and Human Movement, University of Palermo. Centro Forte Feldenkrais di Caterina Forte, Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No